CLINICAL TRIAL: NCT05589948
Title: Radicle™ Calm 1: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Feelings of Anxiety, Stress and Other Health Outcomes
Brief Title: Radicle Calm 1: A Study of Health and Wellness Products on Feelings of Anxiety, Stress and Other Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D04
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo Control 1 (Placebo Comparator): Calm Product Form 1 - control
  Interventions: Dietary Supplement: Radicle Calm Study Placebo Control 1
- Placebo Control 2 (Placebo Comparator): Calm Product Form 2 - control
  Interventions: Dietary Supplement: Radicle Calm Study Placebo Control 2
- Active Product 1.1 (Experimental): Calm Product Form 1 - active product 1
  Interventions: Dietary Supplement: Radicle Calm Study Active Product 1.1
- Active Product 2.1 (Experimental): Calm Product Form 2 - active product 1
  Interventions: Dietary Supplement: Radicle Calm Study Active Product 2.1
- Active Product 2.2 (Experimental): Calm Product Form 2 - active product 2
  Interventions: Dietary Supplement: Radicle Calm Study Active Product 2.2

INTERVENTIONS:
Dietary Supplement: Radicle Calm Study Placebo Control 1 — Participants will use their Radicle Calm Placebo Control Product 1 as directed for a period of 4 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Radicle Calm Study Placebo Control 2 — Participants will use their Radicle Calm Placebo Control Product 2 as directed for a period of 4 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Radicle Calm Study Active Product 1.1 — Participants will use their Radicle Calm Active Product 1.1 as directed for a period of 4 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Radicle Calm Study Active Product 2.1 — Participants will use their Radicle Calm Active Product 2.1 as directed for a period of 4 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Radicle Calm Study Active Product 2.2 — Participants will use their Radicle Calm Active Product 2.2 as directed for a period of 4 weeks.
  Arms: Active Product 2.2

SUMMARY:
A randomized, blinded, placebo-controlled, direct-to-consumer study assessing the impact of health and wellness products on feelings of anxiety, stress and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with up to 300 adult participants per study arm, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for less feelings of anxiety and/or stress, (2) indicate an interest in taking a health and wellness product to potentially improve their anxiety and/or stress, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data will be collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses feelings of anxiety or stress as a primary issue (desire to reduce anxiety or less stress)
* Selects feelings of anxiety/stress, looking to improve their feelings of anxiety/stress, and/or reduce reliance on medications as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid physical shipping address
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Lack of reliable daily access to the internet
* Reports taking anticoagulants, any medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, or MAOIs (monoamine oxidase inhibitors)
* Reports current or recent (within 3 months) use of chemotherapy, immunotherapy, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1211 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in feelings of anxiety | 4 weeks
  Mean difference in feelings of anxiety score as assessed by Patient Reported Outcome Measurement System (PROMIS) Anxiety 8A (scale 8-40; where lower scores correspond to less feelings of anxiety)

SECONDARY OUTCOMES:
Minimal clinically important difference (MCID) in anxiety | 4 weeks
  Likelihood of experiencing a MCID in anxiety score as assessed by PROMIS Anxiety 8A
Change in stress | 4 weeks
  Mean difference in stress score as assessed by PROMIS Stress 8A (scale 8-40; where lower scores correspond to less stress)
Minimal clinically important difference (MCID) in stress | 4 weeks
  Likelihood of experiencing a MCID in stress score as assessed by PROMIS Stress 8A
Change in sleep disturbance | 4 weeks
  Mean difference in sleep disturbance score as assessed by PROMIS Sleep 4A (scale 4-20; where lower scores correspond to better sleep quality/less sleep disturbance)
Change in cognitive function | 4 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognition Function 4A (scale 4-20; where lower scores correspond to poorer cognitive function)

OTHER OUTCOMES:
Change in mood (emotional distress) | 4 weeks
  Mean difference in mood score as assessed by PROMIS Emotional Distress-Depression 4A (scale 4-20; where lower scores correspond to lower levels of emotional distress)
Change in libido | 4 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 4-20; where lower scores correspond to less interest in sexual activity)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com